CLINICAL TRIAL: NCT05345327
Title: SGLT2 Inhibitors As First Line Therapy to Prevent Renal Decline in Type 2 Diabetes
Acronym: START
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The George Institute (Other)
Collaborators: The University of New South Wales (Other); Monash University (Other); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P01148
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Renal decline; Metformin; Sodium Glucose Co-Transporter 2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin 10mg (Experimental): 1x over-encapsulated Dapagliflozin 10mg tablet and 2x Metformin placebo tablets, taken orally once daily for 2 years
  Interventions: Drug: Dapagliflozin
- Metformin XR 2000mg (Active Comparator): 2x Metformin XR 1000mg tablets and 1x over-encapsulated Dapagliflozin placebo, taken orally once daily for 2 years
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Dapagliflozin — SGLT2 inhibitor
  Arms: Dapagliflozin 10mg
Drug: Metformin — Metformin
  Arms: Metformin XR 2000mg

SUMMARY:
The aim of the trial is to evaluate the effects of the SGLT2 inhibitor, dapagliflozin, compared to metformin on annual decline in eGFR when used as first line therapy in people with Type 2 Diabetes.

DETAILED DESCRIPTION:
This study is a randomised, double blinded clinical trial and will be undertaken in primary care and community sites across Australia and tertiary care centres in Sri Lanka. Following a 4-week active run-in period, eligible participants will be randomised to either dapagliflozin 10mg daily, or metformin XR 2000mg daily in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2D;
* Aged ≥18 years;
* Body mass index > 18.5 kg/m2;
* Drug naïve, or managed with metformin monotherapy and willing to be randomised to either dapagliflozin or metformin;
* eGFR ≥45 ml/min/1,73m2; and
* Signed informed consent.

Exclusion Criteria:

* Have an immediate need for rapid intensification of glucose lowering therapy due to marked hyperglycaemia; or
* There is a definite indication for, or contraindication to, either metformin or SGLT2 inhibitor; or
* They have clearly documented coronary artery disease (defined as a previous acute coronary syndrome, coronary stent or bypass surgery) or clearly documented heart failure (defined on the basis of a hospital admission, specialist diagnosis or an echocardiogram or other imaging modality); or
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 994 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of decline in eGFR | 24 months
  Change in estimated glomerular filtration rate (eGFR) from study baseline to 24 months, in ml/min/1.73m2/year

SECONDARY OUTCOMES:
Urine albumin creatinine ratio | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on urine albumin creatinine ratio (mg/g)
Serum creatinine | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on serum creatinine (umol/L)
HbA1C | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on HbA1C (%)
Fasting blood glucose | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on fasting blood glucose (mmol/L)
Systolic and diastolic blood pressure | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on systolic and diastolic blood pressure (mmHg)
Body weight | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on body weight (kg)
Quality of life measured by EQ-5D-5L | 24 months
  Effects of dapagliflozin vs metformin, from baseline to 24 months, on quality of life measured by European Quality of Life 5-Dimensional Assessment, 5-Level version
Anxiety and depression symptoms measured by HADS | 24 months
  Effects of dapagliflozin vs. metformin, from baseline to 24 months, on anxiety and depression symptoms measured by the Hospital Anxiety and Depression Scale (HADS)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Neal, Study Chair — The George Institute for Global Health (Sydney, Australia); Clare Arnott, Study Chair — The George Institute for Global Health (Sydney, Australia)
Locations (8):
- Australia (3):
  - The George Institute for Global Health, Sydney, New South Wales
  - The George Institute for Global Health, Brisbane, Queensland
  - Monash University, Melbourne, Victoria
- Sri Lanka (5):
  - National Hospital - Galle, Galle, Southern Province
  - National Hospital of Sri Lanka 1, Colombo
  - National Hospital of Sri Lanka 2, Colombo
  - Jaffna Teaching Hospital, Jaffna
  - Kandy National Hospital, Kandy

IPD SHARING:
Plan to Share IPD: Yes